CLINICAL TRIAL: NCT05260762
Title: Personalized Obesity Management - Matching Dietary Fibers and Microbial Enterotype (POMFAME)
Brief Title: Personalized Obesity Management - Matching Dietary Fibers and Microbial Enterotype
Acronym: POMFAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Faidon Magkos, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-360
Record Dates: First submitted 2022-01-10; First posted 2022-03-02 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: Gut microbiota; Dietary fiber
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — arabinoxylan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arabinoxylan (Active Comparator): Arabinoxylan (15 g AX/d) wheat buns
  Interventions: Dietary Supplement: Arabinoxylan
- Control (Placebo Comparator): Non-fiber, carbohydrate control (15 g /d) wheat buns
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Arabinoxylan — Dietary fiber product
  Arms: Arabinoxylan
Dietary Supplement: Control — Potato starch
  Arms: Control

SUMMARY:
The overall aim of this 12-week randomized controlled trial is to investigate if a dietary fiber supplement rich in arabinoxylans (AX) affects weight loss success differently according to baseline gut microbiota composition in subjects who have overweight or obesity.

105 participants will be randomized in a 2:1 ratio to receive 15 g/day of AX or placebo.

DETAILED DESCRIPTION:
First, we hypothesize that participants who have a predominantly Prevotella enterotype (inferred by a high Prevotella/Bacteroides-ratio) will lose more body weight after AX supplementation compared to participants with a predominantly Bacteroides enterotype (inferred by a low Prevotella/Bacteroides-ratio). Specifically, we hypothesize that weight loss and P/B-ratio will be positively correlated in the AX supplementation-group whereas there will be no such correlation in the control-group. Consequently, we hypothesize that participants with the Bacteroides enterotype - and the lowest P/B-ratio - will have no benefit after AX supplementation while the weight loss effect of the AX supplementation will increase with increasing P/B-ratio.

Second, we hypothesize that the ability to digest starch in the upper gastrointestinal tract - evaluated by salivary alpha amylase gene (AMY1) copy number - will influence the interactions among AX intake, P/B ratio, and body weight change. Specifically, we hypothesize that there will be an association between body weight change and P/B ratio among subjects with a low AMY1 copy number, but not among the ones with a high AMY1 copy number, when consuming AX.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men or women (self-reported nonpregnant, nonlactating, and not planning a pregnancy in the next 4 months)
* BMI: 25 to 40 kg/m2
* Non-smoker
* Want to maintain or lose weight
* Willing to consume wheat buns on a daily basis

Exclusion Criteria:

* Consumption of whole grain products with every meal
* Use of antibiotics 60 days prior to the start of the study. If a participant uses antibiotics prior to randomization, they will be invited to be re-screened 3 months after the last use of antibiotics, provided that it is realistic to complete the study no later than the scheduled LPLV
* Dietary supplements with pro- and/or prebiotics 6 weeks prior to study
* Self-reported eating disorders
* Being a bodybuilder (>4 strength training sessions per week)
* Alcohol intake above the recommendation from the Danish Health and Medicines Authority (>21 units of alcohol per week)
* Night- or shift work
* Chronic diseases e.g. cancer within the past 5 years (except adequately-treated localized basal cell skin cancer), asthma, thyroid disease, cardiovascular disease, type 1 or 2 diabetes, inflammatory diseases, and celiac disease
* Disorders: neurological, sleep, diagnosed psychiatric disorder and gastrointestinal and liver disorders
* Surgical treatment of obesity and abdominal surgery
* Inability, physically or mental, to comply with the procedures required by the study protocol as evaluated by the daily study manager, principal investigator or clinical responsible
* Subject's general condition contraindicates continuing the study as evaluated by the daily study manager, principal investigator or clinical responsible
* Simultaneous blood donation for another purpose than this study
* Simultaneous participation in other clinical intervention studies

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Body weight change | Baseline to week 12
  Weight will be measured using a calibrated digital scale,in kg to the nearest 0.1 kg

SECONDARY OUTCOMES:
Body fat change | Baseline to week 12
  Evaluated by use of Dual X-ray absorptiometry (DXA) scans
Fecal microbiota composition | Baseline to week 12
  Changes in relative abundance of gut bacteria
Blood glucose metabolism | Baseline to week 12
  Fasting plasma glucose (and insulin) concentrations
Resting energy expenditure | Baseline to week 12
  Indirect calorimetry with canopy mode

OTHER OUTCOMES:
Blood Pressure | Baseline to week 12
  Systolic and diastolic blood pressure and pulse rate will be measured using a validated automatic device on the arm after 5-10 min rest in a resting position.
Blood cholesterol concentration | Baseline to week 12
  Total, LDL and HDL concentrations
Appetite regulating hormones | Baseline to week 12
  ghrelin, glucagon-like peptide-1 (GLP-1), peptide YY (PYY), and cholecystokinin (CCK)
Fecal consistency | Baseline to week 12
  Assessment of fecal consistency by 3-day records
Energy and macronutrient intake | Baseline to week 12
  Assessment of dietary intake by 3-day dietary records
Subjective gastrointestinal (GI) symptoms | Baseline to week 12
  Assessment of subjective GI symptoms via visual analogue scales [1 (low) to 10 (high)]
Subjective appetite sensation | Baseline to week 12
  Assessment of subjective appetite sensation via visual analogue scales [1 (low) to 10 (high)]
Assessment of Brown Adipose Tissue (BAT) activity | Baseline to week 12
  Thermographic camera
Fecal energy concentration | Baseline to week 12
  By bomb calorimeter
Urine metabolome | Baseline to week 12
  Urine metabolome as determined by untargeted metabolic profiling by LC-QTOF of urine samples
Fecal metabolome | Baseline to week 12
  Fecal metabolome as determined by untargeted metabolic profiling by LC-QTOF
Plasma metabolome | Baseline to week 12
  Plasma metabolome as determined by untargeted metabolic profiling by LC-QTOF

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Frederiksberg, Denmark